CLINICAL TRIAL: NCT06521047
Title: A Multicentre Observational Study to Assess Long-term Outcome of Participants in the EXCELLENT Clinical Trial
Acronym: PERFECT
Status: Recruiting | Type: Observational
Sponsor: CellProthera (Industry)
Responsible Party: Sponsor
Other Study IDs: CPT-MI-R01
Record Dates: First submitted 2024-07-09; First posted 2024-07-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Acute Myocardial Infarction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Standard of Care: Patients randomized in the standard of care arm in the EXCELLENT trial who have completed their 6-month follow-up visit
  Interventions: Other: NA - Observational study
- ProtheraCytes Arm: Patients randomized in the ProtheraCytes arm in the EXCELLENT trial, who received an injection of ProtheraCytes and who have completed their 6-month follow-up visit
  Interventions: Other: NA - Observational study

INTERVENTIONS:
Other: NA - Observational study — Observational study, data collection only.

SUMMARY:
The PERFECT study is an observational study designed to follow patients randomised in the EXCELLENT study (NCT02669810) for 10 years.

The aim is to assess the long-term clinical outcomes for patients randomised to the Standard of Care arm or the ProtheraCytes arm.

ELIGIBILITY:
Inclusion criteria :

* Completion of the last visit in the EXCELLENT interventional clinical trial.
* Participation must be within 10 years after the randomization in the EXCELLENT trial

Exclusion criteria :

* Patients randomized to the ProtheraCytes® group who did not receive the product of the EXCELLENT Trial are excluded.
* Any other coexisting conditions that will preclude participation in the study or compromise ability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To be eligible for this observational study, participants must have completed the last visit in the EXCELLENT interventional clinical trial.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2024-07-20 (Actual); Primary Completion 2034-03-15 (Estimated); Study Completion 2034-03-15 (Estimated)

PRIMARY OUTCOMES:
Comparison of the safety and efficacy of patients included in the Protheracytes arm versus the Standard of care arm | Through study completion, an average of 10 year
  The data collected for the efficacity part are cardiovascular markers : NT-Pro-BNP, LVESVI, LVEDVI, LVEF
  The data collected for the safety are : Occurence of Acute Heart failure, Acute MI, transplantation or MACE. All SAE/AE ongoing at or starting from the participant's last visit of the EXCELLENT clinical trial until 10 years after enrolment

CONTACTS AND LOCATIONS:
Locations (10):
- France (6):
  - GHRMSA, Mulhouse, France
  - CHU DIJON Hôpital François Mitterrand 14 rue Gaffarel, Dijon
  - Institut Jacques Cartier, Massy
  - CHU Montpellier Arnaud-De-Villeneuve, Montpellier
  - Hôpital Haut Levèque, Pessac
  - Hôpital de Rangueil, Toulouse
- United Kingdom (4):
  - Ninewells Hospital & Medical School, Dundee
  - BIRMINGHAM, Queen Elizabeth Hospital ,Mindelsohn Way,, Edgbaston
  - University of Edinburgh, Edinburgh
  - Saint Bartholomew's Hospital W Smithfield,, London